CLINICAL TRIAL: NCT01578317
Title: Characterization of Innate Immune Responses to AS03 Adjuvanted H5N1 Vaccine Compared to Non-adjuvanted H5N1 Vaccine
Brief Title: Immune Responses to H5N1 Vaccine With and Without AS03 Adjuvant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 120103; 12-I-0103
Record Dates: First submitted 2012-04-04; First posted 2012-04-16 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-09

CONDITIONS: Influenza
Keywords: H5N1 Vaccine; H5N1 Immunization; AS03 Adjuvant; Biologic Sample Collection; Laboratory Research Specimens; Healthy Volunteer; HV
MeSH Terms: conditions — Influenza, Human | interventions — AS03 adjuvant; Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- AS03 adjuvanted (Experimental): Adminsitered day 1, booster at Day 21
  Interventions: Biological: H5N1 vaccine plus AS03 adjuvant
- unadjuvanted (Experimental): Administer day 1 and booster at Day 21
  Interventions: Biological: H5N1 vaccine without adjuvant

INTERVENTIONS:
Biological: H5N1 vaccine plus AS03 adjuvant — H5N1 influenza vaccine with AS03 at the 3.75 mcg dose level given 21 days apart.
  Arms: AS03 adjuvanted
Biological: H5N1 vaccine without adjuvant — H5N1 influenza vaccine non- adjuvanted form at the 3.75 mcg dose level given 21 days apart.
  Arms: unadjuvanted

SUMMARY:
Background:

- Adjuvants are substances included in vaccines that stimulate the immune system and increase the body's response to the vaccine. The AS03 adjuvant is used in seasonal flu vaccines in Europe. However, it has not been fully tested in the United States. Researchers want to test the immune responses of people who receive a bird flu vaccine with or without AS03 to better understand how the adjuvant works. This information may help develop better flu vaccines.

Objectives:

- To compare the healthy immune system responses to bird flu vaccine with or without the AS03 adjuvant.

Eligibility:

- Healthy volunteers between 18 and 45 years of age.

Design:

* Participants will be screened with a physical exam and medical history.
* Participants will be assigned to one of two groups. Each group will have an initial vaccine, followed by a booster vaccine 21 days later. Both vaccinations will use the same type of vaccine. One group will have the vaccine with AS03; the other group will have the vaccine without it.
* All participants will have two 36-hour inpatient stays to receive the vaccine. Each stay will involve the vaccination, followed by regular and frequent blood draws. Participants will be monitored for any signs or symptoms that may be caused by the vaccine.
* Additional blood samples will be collected 7, 28, 42, and 100 days after the initial vaccination.

DETAILED DESCRIPTION:
Adjuvants have been in use for many decades to enhance the effects of vaccines on the host immune system, yet we know very little on how they actually work. Better understanding of the mechanism by which adjuvants activate the immune system will enable us to develop better and safer vaccines as well as a broad range of immune interventions to a wide spectrum of diseases including cancer and autoimmunity.

In the current study we propose to study the effect of AS03 adjuvant on the innate/early immune response to H5N1, avian flu, a potentially lethal disease that most subjects are assumed to be naive to AS03 is an adjuvant oil in water emulsion containing DL-alpha-tocopherol, squalene and the non-ionic detergent Tween 80 that has been widely used as an adjuvant to flu vaccines produced by GlaxoSmithKline(GSK).

We therefore propose to randomize up to 60 healthy volunteers into two intervention arms (25 volunteers in each arm with up to 10 total replacements in the event a volunteer does not return for the first vaccine). The first arm will receive a vaccine containing H5N1 with AS03 adjuvant, the second arm will receive H5N1 without AS03 adjuvant. Both arms will receive primary and booster vaccination followed by repeated blood sampling to evaluate the immune responses. We will apply high throughput analytic techniques and use systems biology methods to integrate the collected data and draw a description of the immune system response with and without the adjuvant.

The primary objective is to compare multiplex immune response signatures following two (primary and a boost) vaccinations with the GSK AS03 adjuvanted H5N1 influenza vaccine, or the non-adjuvanted form of the H5N1 influenza vaccine, at the 3.75 mcg dose and given 21 days apart and identify differences in very early innate immune responses. These immune signatures will also be correlated with the clinical observations especially safety related local and systemic events.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Healthy status confirmed by History, Physical Exam and blood work through the CHI Screening Protocol.
  2. Age 21 years to 45 years
  3. Able to comprehend the investigational nature of the protocol and provide informed consent
  4. Must be willing to use effective birth control for one month before, during and for two months after the last vaccination.

EXCLUSION CRITERIA:

1. Severe allergies to eggs or their products, chicken proteins or to any component of the influenza antigen preparation.
2. Recipient of AS03 vaccine at any time in the past
3. Recipient of the seasonal influenza vaccine within the past 3 months.
4. Prior severe reactions to vaccines, including influenza vaccines (e.g. anaphylaxis, angioedema or urticaria)
5. Participation on any blood collection or blood donation procedure during study that will bring the total blood draw >550ml over 8 weeks
6. Current pregnancy (women of child bearing potential must have a negative serum pregnancy test done on screening within 1 week of protocol accrual)
7. Currently breast-feeding
8. History of Guillain Barre syndrome
9. Acute illness with patient reported temperature of 38 (Infinite)C or greater within 3 days prior to the proposed time of administration.
10. Any history or presence of serious illness, bleeding disorders or autoimmune disorders, or planned surgeries.
11. Weight less than 50 kg (110 pounds)
12. History of hepatitis or liver disease.
13. Subjects receiving immunosuppressive therapy.
14. Presence of HLA DQB1*06:02, the narcolepsy risk associated allele.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2012-03-20; Primary Completion 2016-01-31 (Actual); Study Completion 2016-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John S Tsang, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Atmar RL, Keitel WA, Patel SM, Katz JM, She D, El Sahly H, Pompey J, Cate TR, Couch RB. Safety and immunogenicity of nonadjuvanted and MF59-adjuvanted influenza A/H9N2 vaccine preparations. Clin Infect Dis. 2006 Nov 1;43(9):1135-42. doi: 10.1086/508174. Epub 2006 Sep 25. PMID 17029131
- [Background] Banzhoff A, Gasparini R, Laghi-Pasini F, Staniscia T, Durando P, Montomoli E, Capecchi PL, di Giovanni P, Sticchi L, Gentile C, Hilbert A, Brauer V, Tilman S, Podda A. MF59-adjuvanted H5N1 vaccine induces immunologic memory and heterotypic antibody responses in non-elderly and elderly adults. PLoS One. 2009;4(2):e4384. doi: 10.1371/journal.pone.0004384. Epub 2009 Feb 6. PMID 19197383
- [Background] Podda A. The adjuvanted influenza vaccines with novel adjuvants: experience with the MF59-adjuvanted vaccine. Vaccine. 2001 Mar 21;19(17-19):2673-80. doi: 10.1016/s0264-410x(00)00499-0. PMID 11257408
- [Result] Khurana S, Coyle EM, Manischewitz J, King LR, Gao J, Germain RN, Schwartzberg PL, Tsang JS, Golding H; and the CHI Consortium. AS03-adjuvanted H5N1 vaccine promotes antibody diversity and affinity maturation, NAI titers, cross-clade H5N1 neutralization, but not H1N1 cross-subtype neutralization. NPJ Vaccines. 2018 Oct 1;3:40. doi: 10.1038/s41541-018-0076-2. eCollection 2018. PMID 30302282
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-I-0103.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AS03 Adjuvanted | Unadjuvanted
Started | 22 | 21
Analysis Population | 22 | 20
Completed | 22 | 20
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AS03 Adjuvanted | Unadjuvanted | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.59 (6.64) | 30.85 (5.62) | 32.28 (6.25)
Sex: Female, Male [Count of Participants; unit: Participants] — self reported
  Participants
    Female | 13 | 12 | 25
    Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Self reported
  Participants
    Hispanic or Latino | 1 | 2 | 3
    Not Hispanic or Latino | 21 | 18 | 39
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Self reported
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 3 | 3
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 6 | 4 | 10
    White | 13 | 12 | 25
    More than one race | 2 | 1 | 3
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Flu Antibody Titers
Description: Flu Antibody titers at days 0, 21, 42, 100. Antibody-neutralization titers by microneutralization were measured against five different H5N1 virus strains (i.e., A/Vietnam/1194/2004 (clade 1), A/Indonesia/5/2005 (clade 2.1), A/Turkey/15/2006 (clade 2.2), A/Egypt/3072/2010 (clade 2.2), and A/Anhui/1/2005 (clade 2.3.4)) at day 0 (prevaccination), day 21 (post first vaccination), day 42 (post second vaccination) and day 100 postvaccination for AS03-adjuvanted group and unadjuvanted group. Sera were tested at an initial dilution of 1:20, and those that were negative (<1:20) were assigned a titer of 10.
Time Frame: Days 0, 21, 42, and 100
Measure: Geometric Mean (Standard Deviation); unit: Titers
Arm/Group | AS03 Adjuvanted | Unadjuvanted
Number analyzed (Participants) | 22 | 20
Titers
  A/Indonesia/5/05 Day 0 | 10.65 (6.4) | 10.35 (2.24)
  A/Indonesia/5/05 Day 21 | 31.09 (60.53) | 10.35 (2.24)
  A/Indonesia/5/05 Day 42 | 600.92 (487.05) | 20 (74.64)
  A/Indonesia/5/05 Day 100 | 218.57 (133.05) | 18.59 (49.14)
  A/Turkey/15/2006 Day 0 | 10.32 (2.13) | 10 (0)
  A/Turkey/15/2006 Day 21 | 10.99 (15.95) | 10 (0)
  A/Turkey/15/2006 Day 42 | 93.65 (313.55) | 10.72 (6.71)
  A/Turkey/15/2006 Day 100 | 34.82 (20.12) | 11.16 (3.75)
  A/Egypt/3072/2010 Day 0 | 10.65 (6.4) | 10 (0)
  A/Egypt/3072/2010 Day 21 | 14.59 (34.83) | 10 (0)
  A/Egypt/3072/2010 Day 42 | 136.68 (291.7) | 11.89 (16.7)
  A/Egypt/3072/2010 Day 100 | 40 (35.02) | 11.57 (9.46)
  A/Anhui/1/2005 Day 0 | 10.65 (6.4) | 10 (0)
  A/Anhui/1/2005 Day 21 | 12.87 (16.77) | 10 (0)
  A/Anhui/1/2005 Day 42 | 106.23 (173.42) | 10.72 (6.71)
  A/Anhui/1/2005 Day 100 | 45.95 (33.78) | 12 (9.55)
  A/Vietnam/1203/2004 Day 0 | 10.65 (6.4) | 10 (0)
  A/Vietnam/1203/2004 Day 21 | 10.99 (14.92) | 10 (0)
  A/Vietnam/1203/2004 Day 42 | 20 (66.76) | 10 (0)
  A/Vietnam/1203/2004 Day 100 | 11.49 (15.69) | 10 (0)

ADVERSE EVENTS:
Arm/Group | AS03 Adjuvanted | Unadjuvanted
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 17/22 | 13/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AS03 Adjuvanted (N=22) | Unadjuvanted (N=20)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Decreased Hemoglobin (Blood and lymphatic system disorders) | 2 (5) | 5 (5)
Decreased Neutrophils (Blood and lymphatic system disorders) | 3 (3) | 3 (4)
Decreased White Blood Cells (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Increased White Blood Cells (Blood and lymphatic system disorders) | 3 (5) | 1 (1)
Fatigue (General disorders) | 3 (4) | 1 (2)
Fever (General disorders) | 7 (7) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 3 (6)
Increased Respiratory Rate (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 4 (8)
Injection Site Redness (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (10) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (6)
Pain at Injection Site (Skin and subcutaneous tissue disorders) | 6 (7) | 1 (1)
Sore Throat (Gastrointestinal disorders) | 3 (3) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes